CLINICAL TRIAL: NCT01603524
Title: Integrating the "Ottawa Model" for Smoking Cessation Into Routine Primary Care Practice: A Cluster Randomized Controlled Trial
Brief Title: Integrating the "Ottawa Model" for Smoking Cessation Into Primary Care Practice
Acronym: RCT-OMSC-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Sophia Papadakis, Program Director, Primary Care Smoking Cessation Program, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011583-01H; NA 7193 (Other Grant/Funding Number: Heart and Stroke Foundation of Canada)
Record Dates: First submitted 2012-05-18; First posted 2012-05-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Smoking Cessation
Keywords: Ottawa Model for Smoking Cessation; Primary Care
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMSC Group (Active Comparator): The OMSC Group will receive a multi-component intervention which includes:
  1. Coaching and Outreach Facilitation Visits: Each practice will receive on-site support to implement the intervention components.
  2. Practice tools and real time prompts: Practices will be provided with 4 tools to support the integration of evidence-based cessation practices into brief clinical encounters as part of a practice-level strategy.
  3. Provider Training in Smoking Cessation Interventions: All clinic providers will be invited to a 3 hour training workshop on smoking cessation(CME).
  4. Telephone follow-up support program: Clinics will be able to refer smokers embarking upon a quit attempt to the smoker's telephone follow-up counseling program.
  Interventions: Other: OMSC Group; Behavioral: OMSC + Performance Feedback Group
- OMSC + Performance Feedback Group (Experimental): The OMSC + Provider Performance Feedback Group will receive the same intervention program as the OMSC group. In addition, clinicians will complete a one-hour audit and feedback session prior to the implementation of the OMSC program at their clinic.
  Interventions: Behavioral: OMSC + Performance Feedback Group

INTERVENTIONS:
Other: OMSC Group — The OMSC Group will receive a multi-component intervention which includes:
  1. Coaching and Outreach Facilitation Visits: Each practice will receive on-site support to implement the intervention components.
  2. Practice tools and real time prompts: Practices will be provided with 4 tools to support the integration of evidence-based cessation practices into brief clinical encounters as part of a practice-level strategy.
  3. Provider Training in Smoking Cessation Interventions: All clinic providers will be invited to a 3 hour training workshop on smoking cessation(CME).
  4. Telephone follow-up support program: Clinics will be able to refer smokers embarking upon a quit attempt to the smoker's telephone follow-up counseling program.
  Arms: OMSC Group
Behavioral: OMSC + Performance Feedback Group — The OMSC + Performance Feedback Group will receive the same intervention program as the OMSC group. In addition, clinicians will complete a one-hour audit and feedback session prior to the implementation of the OMSC program at their clinic. The goal of the audit and feedback is to increase provider self-efficacy in the delivery of smoking cessation interventions, raise awareness of the current delivery of evidence-based cessation practices, identify areas for improvement, and motivate providers to deliver evidence-based treatments.

SUMMARY:
This proposal outlines the design of a cluster randomized controlled trial to compare the effectiveness of a new approach to integrating smoking cessation services into routine interactions with patients in the primary care setting using an adaptation of the Ottawa Model for Smoking Cessation (OMSC). The OMSC aims to systematically identify the smoking status of all patients, provide brief cessation advice, and offer evidence-based cessation support to those interested in embarking on a quit attempt. This study will provide important new evidence to assist with the development of a more comprehensive cessation system in the province of Ontario and across Canada.

DETAILED DESCRIPTION:
A multi-component intervention has been designed to facilitate the uptake of the OMSC using best evidence regarding the integration of smoking cessation intervention into primary care practice. The secondary objective of the study is to examine the incremental value of providing tailored performance feedback to primary care practitioners when delivered as part of the OMSC intervention program.

ELIGIBILITY:
Practice Inclusion Criteria:

* Is a primary care practice (family health team, family health group, family health network, community health centre);
* Has a minimum of five full time physicians on staff or sees an average of 50 patients per day;
* All physicians within the practice are willing to participate in the study.

Practice Exclusion Criteria:

* Primary care practices with less than 5 family physicians in a shared clinic space will be excluded.
* Clinics who have already implemented the OMSC will also be excluded.

Patient Inclusion Criteria:

* Current smoker (>5 cigarette per day on most days of the week);
* 18 years of age or older;
* Scheduled for an annual exam or non-urgent medical appointment with a physician or nurse practitioner;
* Able to read and understand English or French;
* Has a home or mobile telephone which can be used to receive follow-up telephone counselling calls;
* Has the mental capacity to provide informed consent and complete study protocols.

Patient Exclusion Criteria:

* Unable to read and understand English or French;
* Do not have a home or mobile telephone which can be used to receive follow-up calls;
* Do not have the mental capacity to provide informed consent and complete study protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Effect of the Ottawa Model for Smoking Cessation within family doctors' offices compared to control practices. | Patient bio-chemically verified 7-day point prevalence abstinence is measured at 6 months post-enrollement.
  The primary objectives of this study are to determine whether the Ottawa Model for Smoking Cessation (OMSC) increases:
  1. the delivery of evidence-based smoking cessation interventions within family doctors' offices,
  2. number of patient quit attempts, and
  3. patient bio-chemically verified 7-day point prevalence abstinence measured at 6-months compared to standard care control practices.

SECONDARY OUTCOMES:
Examining the incremental impact of audit and feedback within family doctors' offices compared to the OMSC alone group and standard control practices. | Patient bio-chemically verified 7-day point prevalence abstinence is measured at 6 months post-enrollement.
  The secondary objectives of this study are to examine the incremental impact of audit and feedback on:
  1. provider delivery of evidence-based smoking cessation interventions,
  2. number of patient quit attempts, and
  3. 7-day point prevalence abstinence measured at 6-months in family doctors' offices compared to the OMSC alone and standard care control practices.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Papadakis, Ph.D., MHA, Principal Investigator — University of Ottawa Heart Insitute; Andrew Pipe, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Reid RD, Mullen KA, Slovinec D'Angelo ME, Aitken DA, Papadakis S, Haley PM, McLaughlin CA, Pipe AL. Smoking cessation for hospitalized smokers: an evaluation of the "Ottawa Model". Nicotine Tob Res. 2010 Jan;12(1):11-8. doi: 10.1093/ntr/ntp165. Epub 2009 Nov 10. PMID 19903737
- [Background] Papadakis S, McDonald P, Mullen KA, Reid R, Skulsky K, Pipe A. Strategies to increase the delivery of smoking cessation treatments in primary care settings: a systematic review and meta-analysis. Prev Med. 2010 Sep-Oct;51(3-4):199-213. doi: 10.1016/j.ypmed.2010.06.007. Epub 2010 Jun 17. PMID 20600264
- [Background] McIvor A, Kayser J, Assaad JM, Brosky G, Demarest P, Desmarais P, Hampson C, Khara M, Pathammavong R, Weinberg R. Best practices for smoking cessation interventions in primary care. Can Respir J. 2009 Jul-Aug;16(4):129-34. doi: 10.1155/2009/412385. PMID 19707607
- [Derived] Papadakis S, Pipe AL, Reid RD, Tulloch H, Mullen KA, Assi R, Cole AG, Wells G. Effectiveness of performance coaching for enhancing rates of smoking cessation treatment delivery by primary care providers: Study protocol for a cluster randomized controlled trial. Contemp Clin Trials. 2015 Nov;45(Pt B):184-190. doi: 10.1016/j.cct.2015.08.013. Epub 2015 Sep 5. PMID 26348788